CLINICAL TRIAL: NCT02400008
Title: Selective Bilateral Laryngeal Reinnervation as a Secondary Treatment in Case of Bilateral Vocal Fold Paralysis: Analysis of Phonatory and Ventilatory Results
Brief Title: Selective Bilateral Laryngeal Reinnervation as a Secondary Treatment in Case of Bilateral Vocal Fold Paralysis
Acronym: SEQLAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011/120/HP
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Bilateral Vocal Fold Paralysis
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient with bilateral vocal fold paralysis (Experimental): Patient with bilateral vocal fold paralysis in a closure position between 6 months to 36 months before et who has been treated by endoscopic treatment without satisfying result (voice or breathing).
  Interventions: Procedure: Surgery for bilateral laryngeal reinnervation

INTERVENTIONS:
Procedure: Surgery for bilateral laryngeal reinnervation — Surgery for bilateral laryngeal reinnervation assessed for patient with bilateral vocal fold paralysis

SUMMARY:
Selective laryngeal bilateral reinnervation as a secondary treatment in patients with bilateral vocal fold paralysis, previously treated by endoscopy, without residual arytenoids ankylosis.

The surgical procedure is : functional reinnervation with the upper root of one phrenic nerve, is used for reinnervation of both cricoarytenoid muscles (laryngeal inspiratory muscles), and simultaneous reinnervation of adductor laryngeal muscles is performed by right and left thyro -hyoid nerves (coming from the hypoglossi) on both sides.

Results are obtained after 6 to 9 months delay. In case of good inspiratory arytenoid abduction, and residual dysphonia, a secondary vocal fold medialization is done by an endoscopic approach 12 months after reinnervation (included in the protocol).

Improvement is expected in voice and breathing, without aspiration.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Bilateral vocal fold paralysis in a closure position 6 months to 36 months before.
* Patient who has been treated by endoscopic treatment without satisfying result (voice or breathing).
* Patient with passive mobile arytenoid at least on one side
* Tracheostomized or not
* Age > 18 years old
* Good general situation

Exclusion Criteria:

* Long term vocal fold paralysis (more than 3 years with strong denervation)
* Ary-cricoid ankylosis or synechiae
* Age >75 years
* Anaesthesiologist contra indication
* Strong respiratory disease history
* Severe coagulation troubles
* Ongoing neoplasia disease
* Cardiac pace maker
* Pregnant woman or without contraception
* Impairment of the freedom

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-11-09 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Maximal phonation time | 18 Months
  Maximal phonation time will be assessed at 18 Months

SECONDARY OUTCOMES:
Voice quality assessed using quality of life questionnaire | 18 Months
  Voice quality will be assessed using quality of life questionnaire, computerized analysis, swallowing scores
Voice quality assessed using computerized analysis | 18 Months
  Voice quality will be assessed using computerized analysis
Voice quality assessed using swallowing scores | 18 Months
  Voice quality will be assessed using swallowing scores

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul MARIE, Pr, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France